CLINICAL TRIAL: NCT01776658
Title: Pilot Study to Evaluate SYL1001 Safety and Effect in Patients With Ocular Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sylentis, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYL1001_II
Record Dates: First submitted 2012-11-14; First posted 2013-01-28 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Ocular Pain; Dry Eye Syndrome
Keywords: Ocular pain; Dry Eye Syndrome; siRNA; RNAi; TRPV1
MeSH Terms: conditions — Eye Pain; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- SYL1001 eye drops dose A (Experimental): Ocular topical administration of SYL1001 eye drops dose A
  Interventions: Drug: SYL1001
- Placebo (Placebo Comparator): Ocular topical administration of placebo eye drops
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYL1001 — Ocular topical administration of SYL1001 for 10 consecutive days
  Arms: SYL1001 eye drops dose A
Drug: Placebo — Ocular topical administration of placebo for 10 consecutive days
  Arms: Placebo

SUMMARY:
The aim of this pilot study is to compare the analgesic effect of SYL1001 versus placebo in patients with ocular pain associated with Dry Eye Syndrome. General and local tolerability are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders
* Age ≥ 18 years old
* Give written informed consent to participate in the study after having been informed of the study design, objectives and possible derived risks
* Common mild to moderate dry eye symptoms. Persistent daily symptoms for more than three months:
* OSDI scale: 13-30
* VAS scale: 2-7
* Ocular tests in both eyes:
* Corneal staining with fluorescein. Oxford scale > 0
* Tear Breakup Time Test: (BUT) < 10 seconds
* Schirmer test with anaesthesia < 10 mm/5min

Exclusion Criteria:

* Pregnant or breastfeeding females or those with a positive pregnancy test.
* Females of childbearing potential who will not use a medically acceptable contraceptive method from selection and during the whole study.
* Current relevant disease, including respiratory disease, cardiovascular, endocrine, neurological, haematological, renal, neoplasic, hepatopathy, gastrointestinal distress, hypertension, or infectious acute processes.
* Past history of a chronic o recurring condition that could interfere with study according to the investigator's judgement.
* Concomitant use of other drugs with analgesic activity by any route of administration at the enrolment period.
* Changes in any ocular and/or systemic concomitant medication one month prior to the study commencement and during the study development.
* Changes on the preestablished artificial tears dosage 15 days prior to the study commencement and during the study development.
* Cyclosporine treatment initiation or changes in cyclosporine dosage or dosing regimen during the 6 months prior to enrolment.
* Previous history of drug hypersensitivity.
* Use of contact lenses
* Case history of drug or alcohol abuse or dependence.
* Relevant abnormal laboratory results as judged by the investigator
* Previous refractive surgery
* Participation in a clinical trial within 2 months before the enrolment visit
* Relevant ocular pathology judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline in the Ocular Pain Scores on the Visual Analog Scale (VAS) and in the Ocular Discomfort Scores on the Ocular Surface Disease Index (OSDI) as a Measure of SYL1001 Analgesic Effect versus Placebo. | 10 days + (4-10 days)
Simple Corneal and Conjunctival Evaluation as a Measure of Safety and Tolerability using Ophthalmic Dyes and a Slit Lamp | 10 days + (4-10 days)

SECONDARY OUTCOMES:
Assessment of Adverse Events Appearance as a measure of SYL1001 tolerability | 10 days + (96-240 hours)
Evaluation of Vital Signs, Blood, Urine and Ocular Parameters Alterations (IOP, Visual Acuity, Anterior Segment Exploration) Possibly Related to the Investigational Product | 10 days + (96-240 hours)

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Instituto Oftalmológico Fernández-Vega, Oviedo

REFERENCES:
- [Derived] Benitez-Del-Castillo JM, Moreno-Montanes J, Jimenez-Alfaro I, Munoz-Negrete FJ, Turman K, Palumaa K, Sadaba B, Gonzalez MV, Ruz V, Vargas B, Paneda C, Martinez T, Bleau AM, Jimenez AI. Safety and Efficacy Clinical Trials for SYL1001, a Novel Short Interfering RNA for the Treatment of Dry Eye Disease. Invest Ophthalmol Vis Sci. 2016 Nov 1;57(14):6447-6454. doi: 10.1167/iovs.16-20303. PMID 27893109